CLINICAL TRIAL: NCT04838691
Title: The Effect of Interpersonal Counseling in Symptoms Management of Premenstrual Syndrome
Brief Title: Premenstrual Syndrome and Interpersonal Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Zeynep Seyyide Bozkurt, Principle Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: zeynep
Record Dates: First submitted 2021-04-03; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Premenstrual Syndrome
Keywords: premenstrual syndrome; interpersonal counseling
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interpersonal relations counseling applied (Experimental): 8 sessions of interpersonal relations counseling, each lasting 40 minutes, were applied for 2.
  Interventions: Behavioral: interpersonal counseling
- no application (No Intervention): No action taken.

INTERVENTIONS:
Behavioral: interpersonal counseling — In the intervention group, it will be administered for 40 minutes for 8 weeks to people with symptoms of premenstrual syndrome.
  Arms: interpersonal relations counseling applied

SUMMARY:
This study aims to test the effectiveness of interpersonal counseling in PMS symptom management in university students experiencing PMS symptoms.

DETAILED DESCRIPTION:
People diagnosed with Premestrual Syndrome were identified through an online questionnaire. 80 people who were identified and accepted to study were divided into two groups as experiment and control. Initially, pre-menstrual screening tool, interpersonal relationship dimensions scale and perceived stress scale were applied to all groups. Then, 8 sessions of interpersonal counseling, each lasting 40 minutes, were applied to the experimental group for 2 months. Scales were repeated for both groups after the application was completed. Repeated measurements were made 3 months later.

ELIGIBILITY:
Inclusion Criteria:

1. According to the Pre-menstrual Symptom Screening Instrument, which is located in the group living with AES (Pre-Mental Syndrome)
2. between the ages of 18-30
3. Menstruating at regular intervals for at least 2 years (21-35 days)
4. Those who have never given birth
5. Speak and understand Turkish
6. It will consist of people who have not received antidepressant, oral contraceptive or hormone therapy for any reason.

Exclusion Criteria:

1. Having a known gynecological disease (endometriosis, polycystic ovary, ...)
2. A known, ongoing physical health problem (diabetes, rheumatic disease, ...)
3. Any psychiatric disease diagnosed (psychotic disorder, mood disorder, anxiety disorder ...)
4. People who use cigarettes, alcohol or substances

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women
Enrollment: 80 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Premenstrual Symptom Screening Tool | Baseline (beginning), Change from Baseline PMDD or PMS after 2 months, Change from Baseline PMDD or PMS after 5 months,
  Women will be divided into 3 different groups as a result of the points they get from PSST. The first group will consist of women who fully meet the PMDD criteria. These Women must have at least one of the four main symptom groups from the group A symptoms plus any of the 4 symptoms marked as moderate to severe on the instrument. In addition, he should have reported that at least one of the questions in group B was severe, and yes answers should be given to both questions in group C.The second group is the group that meets the PMS living criteria. These women are expected to have marked at least one of the 4 main symptoms as moderate to severe from the group A questions and any other 4 symptoms as moderate to severe to answer the group B questions as moderate to severe, and to answer yes to at least one question from the C group.The third group will be considered as the group with subthreshold symptoms consisting of those who do not meet the criteria for entering the other two groups.

SECONDARY OUTCOMES:
Scale Of Interpersonal Relatıonshıps Dımensıons | Baseline (beginning), Change from Baseline Sub-dimensions of Interpersonal Relationships Scale after 2 months, Change from Baseline Sub-dimensions of Interpersonal Relationships Scale after 5 months
  The scale, which consists of 53 items in total, has 4 sub-dimensions. These are Confirmation, addiction, empathy, trust in others, and emotional awareness.
  The high score obtained from each sub-dimension of the scale indicates that the individual has more features evaluated by the relevant sub-dimension.
Perceived stress scale | Baseline (beginning), 2 months after beginning, 3 months after beginning
  The higher the total score, the more negative it is.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Özcan, Professor, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing is considered inappropriate before the end of the study.